CLINICAL TRIAL: NCT06814990
Title: Erfassung Kardialer Funktionsparameter in MRT Und Echokardiographie Bei Patienten Mit Ethyltoxischer Leberzirrhose Und Transjugulärer Intrahepatischer Portosystemischer Shunt (TIPSS)-Anlage
Brief Title: Acquisition of Cardiac Function Parameters in MRI and Echocardiography in Patients with Ethyltoxic Liver Cirrhosis and Transjugular Intrahepatic Portosystemic Shunt (TIPSS) Placement
Acronym: EVALUATION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stephanie Gräger (Other)
Collaborators: Jena University Hospital (Other)
Responsible Party: Sponsor-Investigator, Stephanie Gräger, Radiologist, Jena University Hospital
Organization: Jena University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-3204-BO
Record Dates: First submitted 2024-11-13; First posted 2025-02-07 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: MASLD; Liver Cirrhosis, Alcoholic; Cirrhosis of Liver; Heart Decompensation; TIPS
Keywords: Chirrotic cardiomyopathy; Liver chirrosis; TIPS
MeSH Terms: conditions — Liver Cirrhosis, Alcoholic; Fibrosis; Heart Failure | interventions — Blood Specimen Collection; Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Measurements of cardiac function in MRI and echocardiography, additional laboratory work (Experimental): Patients in this arm will receive three additional cardiac magnetic resonance imaging (MRI) scans with acquisition of cardiac function parameters, T1 and T2 relaxation time measurements and a newly introduced 4D-Flow sequence to assess changes in aortic and pulmonary artery flow. These patients will also receive extended echocardiography with additional parameters to diagnose cirrhotic cardiomyopathy. We will also analyse specific blood parameters that are not yet part of the clinical standard.
  Interventions: Diagnostic Test: Cardiac MRI; Diagnostic Test: Blood samples; Diagnostic Test: Echocardiography

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — Additional to standard clinical practice Patients will receive a cardiac magnetic resonance imaging without contrast. Measured parameters are enddoastolic and endsystolic volume (in ml oder ml/body surface area (BSA)), stroke volume (in ml) of right and left ventricle absolute and relatvie to body surface area (BSA), ejection fraction in % of right and left ventricle, myocardial Strain in % of right and left ventricle if applicable. T1 and T2 relaxation times are obtained and aortic and pulmonary artery flow parameters are measured.
Diagnostic Test: Blood samples — We will take additional blood samples for the analysis of markers of bacterial translocation (e.g. LBP, EndoCAb, 16S rRNA), detection of bacterial markers (bacterial extracellular vesicles), inflammatory markers (e.g. IL-1ß, TNF-α, TGF-ß, IL-6, CXCL8, IL1-RA, IL-10, IL-18) and monocyte/macrophage activation markers (sCD14, sCD163, sCD87, sCD206), bile acids (including TCA, GCA, GCDCA, TCDCA, TLCA, GLCA, TDCA, GDCA, CA, CDCA, UDCA, DCA, TUDCA, LCA), lipids and lipoproteins (triglyerides, cholesterol, LDL/HDL cholesterol), coagulation factors (e.g. VWF, ADAMTS13, fibrinogen), markers of cardiac remodeling (e.g. NT-proBNP; troponin, VEGF-D, cleaved Gasdermin D, HMGB1) and Immunophenotyping of monocytes/macrophages, T and B cells (e.g. CD14, CD16, MERTK, CD4, CD127, CD25, TREM1/2).
Diagnostic Test: Echocardiography — Patients will receive an extended echocardiographic protocol. In addition to standard clinical parameters, we will collect study specific parameters such as LV EF in %, global longitudinal strain in %, septal e' velocity (cm/s), E/e' ratio, left atrial volume index (LAVI) (in ml/m2), tricuspid regurgitation velocities (m/s).

SUMMARY:
The aim of this clinical trial is to investigate the development of cardiac decompensation following transjugular intrahepatic portosystemic shunt (TIPSS) implantation in order to draw conclusions for future treatment methods or exclusion criteria prior to TIPS implantation.

The main questions to be answered are:

How often do symptoms of cardiac decompensation develop over a one year period? What laboratory, clinical or imaging morphological changes are associated with this? In addition to the standardised clinical procedure for TIPSS implantation, participants will undergo 3 cardiac magnetic resonance imaging (MRI), extended echocardiographic examinations (both just before, 3 days after and 3 months after implantation) and laboratory chemistry tests for specific endothelial and inflammatory markers (just before, on the day of implantation, 1 day after, 1, 3, 6 and 12 months after implantation).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 99 years
* Written informed consent of the patient
* Decompensated liver cirrhosis, defined by clinical, imaging or laboratory criteria
* Patient receives an elective TIPSS in the appropriate clinical context at the JUH

Exclusion Criteria:

* Pregnancy
* Implants not suitable for magnetic resonance imaging
* Medical/personal reasons against magnetic resonance imaging (claustrophobia, patient cannot lie flat or follow breathing commands)
* Patient in critical condition or incompliant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2027-04-19 (Estimated); Study Completion 2027-04-19 (Estimated)

PRIMARY OUTCOMES:
Determination of the frequency of occurrence of cardiac decompensation | From TIPSS to cardiac decompensation 12 Month
  Cardiac decompensation is defined as one or a collection of the following new symptoms: Fatigue, Dyspnoea, Edema, jugular vein congestion, elevated pro-BNP, restricted heart function in echocardiography, clinically indicated chest x-ray with edema or pleura effusion. Clinical evaluation and diagnostic methods according to clinical standard are applied (e.g. x-ray and ultrasound if clinically needed).

SECONDARY OUTCOMES:
Acquisition of right and left heart function parameters in patients before TIPS implantation | 1day before TIPS-Implantation
  Monitoring changes in cardiac function using cardiac MRI. Measured parameters are end diastolic and end systolic volumes (in ml or ml/BSA), stroke volume (in ml) of the right and left ventricle absolute and relative to body surface area (BSA), ejection fraction in percent of the right and left ventricle, myocardial strain in percent of the right and left ventricle if applicable.
Acquisition of right and left heart function parameters in patients after TIPS implantation | 1-3 days after TIPS-Implantation
  Monitoring changes in cardiac function using cardiac MRI. Measured parameters are end diastolic and end systolic volumes (in ml or ml/BSA), stroke volume (in ml) of the right and left ventricle absolute and relative to body surface area (BSA), ejection fraction in percent of the right and left ventricle, myocardial strain in percent of the right and left ventricle if applicable.
Acquisition of right and left heart function parameters in patients 3 Month after TIPS implantation | about 3 month after TIPS-Implantation
  Monitoring changes in cardiac function using cardiac MRI. Measured parameters are end diastolic and end systolic volumes (in ml or ml/BSA), stroke volume (in ml) of the right and left ventricle absolute and relative to body surface area (BSA), ejection fraction in percent of the right and left ventricle, myocardial strain in percent of the right and left ventricle if applicable.
Acquisition of T1 and T2 mapping without contrast agent administration during the course | 1day before TIPS-Implantation to about 3 Month after
  Detection of changes in T1 and T2-relaxation time in ms in MRI
Evaluation of changes in flow parameters in the aorta and pulmonary artery | 1day before TIPS-Implantation to about 3 Month after
  Using newly implemented 4D Flow in MRI to observe changes in arterial flow and improve clinical usability of the sequence.
Follow-up of echocardiographic parameters and correlation with cardiac MRI | 1day before TIPS-Implantation to about 3 Month after
  Observation of changes in cardiac function via echocardiography and subsequent comparison with cardiac MRI parameters
Correlation with laboratory markers (for inflammation, liver fibrosis, metabolism, cardiac remodeling) | 1day before TIPS-Implantation to about 6 Month after
  Correlation of clinical and imaging parameters with different blood markers which are aquired to clinical standard (Serum sodium, Quick, INR, pTT, Crea, urea, albumin, CRP, ALAT, ASAT, Bili, venous pH, LDH, lactate, glucose, complete blood count) and study specific (markers of bacterial translocation (e.g. LBP, EndoCAb, 16S rRNA), detection of bacterial markers (bacterial extracellular vesicles), inflammatory markers (e.g. IL-1ß, TNF-α, TGF-ß, IL-6, CXCL8, IL1-RA, IL-10, IL-18) and monocyte/macrophage activation markers (sCD14, sCD163, sCD87, sCD206), bile acids (including TCA, GCA, GCDCA, TCDCA, TLCA, GLCA, TDCA, GDCA, CA, CDCA, UDCA, DCA, TUDCA, LCA), lipids and lipoproteins (triglyerides, cholesterol, LDL/HDL cholesterol), coagulation factors (e.g. VWF, ADAMTS13, fibrinogen), markers of cardiac remodeling (e.g. NT-proBNP; troponin, VEGF-D, cleaved Gasdermin D, HMGB1) and Immunophenotyping of monocytes/macrophages, T and B cells (e.g. CD14, CD16, MERTK, CD4, CD127, CD25, TREM1/2).

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Gräger, Principal Investigator — Jena University Hospital; Stefanie Quickert, Principal Investigator — Jena University Hospital; René Aschenbach, Principal Investigator — Jena University Hospital; Alexander Zipprich, Principal Investigator — Jena University Hospital
Locations (1):
- Jena University Hospital, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No